CLINICAL TRIAL: NCT04836299
Title: Randomized, Double-blind, Placebo-controlled Clinical Trial to Study the Efficacy and Therapeutic Safety of Ivermectin Versus Placebo Associated With Standard of Care Treatment in the Early Phase of Coronavirus Infection (COVID19).
Brief Title: Clinical Trial to "Study the Efficacy and Therapeutic Safety of Ivermectin: (SAINTBO)
Acronym: SAINTBO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Mayor de San Simón (Other)
Collaborators: Barcelona Institute for Global Health (Other); Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Jorge Luis Aviles, MD. MPH. PhDc., Universidad Mayor de San Simón
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCT01
Record Dates: First submitted 2021-03-02; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Covid19
Keywords: Efficacy; Safety; Ivermectin
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, Placebo-controlled parallel clinical trial to "Study the efficacy and therapeutic safety of Ivermectin associated with standard of care treatment versus placebo with standard of care treatment in the early phase of coronavirus infection (COVID19).
  A PHASE II pilot study.
Who Masked: Participant, Care Provider
Masking Description: The participants, care providers and also investigator will be blinded for this study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ivermectin (Experimental): Participants will receive a single 600 µg / kg dose of ivermectin.
  Interventions: Drug: Ivermectin
- Placebo Comparator (Placebo Comparator): Participants will receive a single dose of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivermectin — Participants will be randomly assigned to receive a single 600 µg / kg dose of ivermectin or placebo.
  Other Names: A
  Arms: Ivermectin
Drug: Placebo — Participants will be randomly assigned to receive a single of placebo.
  Other Names: B
  Arms: Placebo Comparator

SUMMARY:
Coronavirus disease (COVID-19) is an infectious disease caused by a new virus. The disease causes a respiratory illness (such as the flu) with symptoms such as cough, fever, and, in more severe cases, respiratory distress, even developing Acute Respiratory Distress Syndrome, evolving in some cases with the death of the patient. Currently, there are no specific treatments for COVID-19. Currently, there are several ongoing clinical trials evaluating possible treatments. Recently, Leon Caly reports here that Ivermectin, an FDA-approved antiparasitic that was shown to have broad-spectrum antiviral activity in vitro, is an inhibitor of the causative virus (SARS-CoV-2), with a single addition to Vero cells. hours after infection with SARS-CoV-2 capable of a 5000-fold reduction in viral RNA at 48 h. (1) Ivermectin, therefore, warrants further investigation for possible benefits in humans. The reason for this study is to understand the effect of the drug in eradicating the virus.

It is a randomized controlled trial to evaluate the efficacy of Ivermectin in COVID-19. The recruited patient will be assigned to two groups, (1) a group received ivermectin plus care treatment (2) the placebo group plus standard care treatment. The result will be recorded by documenting the RT-PCR reports confirmed at the time of recruitment and at 7 and 14 days within the framework of the study, then they will be adapted to the national care protocol, with 9 scheduled clinical and telemedicine interviews.

It will be a randomized controlled trial to be run in RT-PCR confirmed COVID-19 patients who meet the inclusion criteria (asymptomatic/mild to moderate severity).

They will be divided into groups after randomization. Group A will be administered one (1) a group received ivermectin plus standard of care treatment (2) the placebo group plus standard of care treatment, along with the existing inpatient and outpatient management clinical guidelines of the hospitals participating in the study, these being adapted to the National standard.

The reverse transcriptase-polymerase chain reaction (RT-PCR) will be carried out on days 7 and 14 after the therapeutic intervention and the duration of time at which the RT-PCR becomes negative and/or clinical evolution of the patient will be compared in both study groups. The dose of the drug is not subject to change according to the patient's response or the possible side effect of being administered in a single dose.

DETAILED DESCRIPTION:
STUDY DESIGN It is a double-blind, randomized, placebo-controlled superiority trial with two parallel arms. Participants will be randomized to receive a single 600 µg / kg dose of ivermectin or placebo, and the number of patients in the treatment and placebo groups will be in a 2: 1 ratio for the intervention group.

The trial statistician will generate the randomization code using blocks of four individuals to ensure the balance between groups. The assignment will be carried out by the main investigator using opaque envelopes, after obtaining informed consent and verification of compliance with all the inclusion and exclusion criteria. The investigational product will be administered by personnel who are not involved in patient care or monitoring of study participants.

Participants will be followed up at their homes for a period of 28 days. A patient can discontinue her participation in the study at any time and for any reason. The principal investigator and the panel of experts that make up the safety and adverse effects committee may also withdraw a patient from the study if they believe it is in the best interest of the patient.

Serious adverse events (SAEs) related to ivermectin will be followed until they resolve or up to 28 days after the participant's final visit, whichever occurs first. All other SAEs deemed unrelated to ivermectin will be followed up until the participant's final visit or for a specified period at the discretion of the principal investigator.

The study will end when the final randomized patient has completed the study, all planned visits have been completed, and inconsistencies in the data have been resolved.

OBJECTIVES Primary objective

• To explore the efficacy and therapeutic safety of Ivermectin in patients with non-severe and low-risk COVID-19 in the first 72 hours after the onset of symptoms, through the negativization of the polymerase chain in real time. RT-PCR (nasopharyngeal swab) and clinical improvement on day 7 and 28 after treatment, to explore its possible use in the fight against the pandemic.

Secondary objectives

1. To evaluate the efficacy of ivermectin in reducing the SARS-CoV-2 viral load in the nasopharyngeal swab on day 7 after treatment.
2. To evaluate the efficacy of ivermectin in improving the progression of symptoms in treated patients.
3. Assess the proportion of seroconversions in patients treated on day 21.
4. Evaluate the safety of ivermectin at the proposed dose.
5. Determine the magnitude of the immune response against SARS-CoV-2
6. Evaluate the early kinetics of immunity against SARS-CoV-2

ELIGIBILITY:
Inclusion Criteria:

* Confirmed case of COVID-19 in national reference hospitals - COVID sentinel hospitals.
* Male and female patients 18 to 75 years (inclusive) of age.
* Supply of signed and dated informed consent form
* Declared availability to comply with all study procedures and availability for the duration of the study.
* In good general health with mild or moderate symptoms during the first week of disease evolution (onset of symptoms maximum 7 days before recruitment).
* Ability to take oral medications and be willing to adhere to the medication consumption regimen prescribed in the study.
* The patient must, in the opinion of the principal investigator, be able to comply with all the requirements of the clinical trial (including home monitoring during isolation).
* The patient is able and willing to comply with the requirements of this test protocol. Voluntarily signed informed consent obtained prior to any proceeding related to the trial.

Exclusion Criteria:

1. Known history of ivermectin allergy
2. Hypersensitivity to any component of ivermectin or the excipients of the brand to be used.
3. COVID-19 pneumonia

   * Diagnosed by the treating physician
   * Identified on a chest x-ray
4. Fever or cough present for more than 48 hours.
5. immunoglobulin G (IgG) positive against SARS-CoV-2 by a rapid diagnostic test

8. Recent travel history to loa endemic countries (Angola, Cameroon, Central African Republic, Chad, the Democratic Republic of the Congo, Ethiopia, Equatorial Guinea, Gabon, Republic of the Congo, Nigeria, and Sudan) 9. Current use of quinidine, amiodarone, diltiazem, spironolactone, verapamil, clarithromycin, erythromycin, itraconazole, ketoconazole, cyclosporine, tacrolimus, indinavir, ritonavir, or cobicistat. Use of critical drugs such as warfarin.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-05-08 (Estimated); Primary Completion 2021-07-08 (Estimated); Study Completion 2021-12-05 (Estimated)

PRIMARY OUTCOMES:
Evolution of viral load | 3 days
  A comparison will be made between the initial viral load before the dose of ivermectin with respect to the viral load on the third day after the administration of the drug. The primary outcome of interest will be the correlation between the use of a treatment regimen containing Ivermectin plus the standard of care, with the endpoint of measurement relative to the difference in viral loads.
Clinical remission | 28 days
  Clinical remission, defined as a remission of all the patient's symptoms based on the clinical management protocol. The primary outcome of interest will be the correlation between the use of a treatment regimen containing Ivermectin plus the standard of care, initiated early after the confirmed diagnosis of COVID-19 with the endpoint of measurement relative to the difference in clinical evolution.

SECONDARY OUTCOMES:
Clinical signs of toxicity | 28 days
  The secondary outcome of interest will be the correlation between these treatment regimens and the appearance of clinical signs of toxicity or adverse effects (defined as the first clinical or laboratory finding of a neurological, hepatic, renal, hematological, or pancreatic alteration, or verification of alterations in pupillometry during the outpatient clinical course or hospitalization.

OTHER OUTCOMES:
Need for supplemental oxygen | 28 days
  The need for supplemental oxygen implementation will be evaluated
Hospital stay | 3 months
  The need for hospital care and the stay both in general wards and in intensive care (ICU) will be evaluated.
Need for mechanical ventilation | 21 days
  The need to implement the intervention through mechanical ventilation will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos L Erostegui, MPH, Study Director — Universidad Mayor de San Simón
Locations (1):
- Universidad Mayor de San Simón, Cochabamba, Bolivia

IPD SHARING:
Plan to Share IPD: Yes
It is planned to grant the respective information stored in a repository.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: until August 2021
Access Criteria: unrestricted access

REFERENCES:
- [Background] Heidary F, Gharebaghi R. Ivermectin: a systematic review from antiviral effects to COVID-19 complementary regimen. J Antibiot (Tokyo). 2020 Sep;73(9):593-602. doi: 10.1038/s41429-020-0336-z. Epub 2020 Jun 12. PMID 32533071
- [Background] Choudhary R, Sharma AK. Potential use of hydroxychloroquine, ivermectin and azithromycin drugs in fighting COVID-19: trends, scope and relevance. New Microbes New Infect. 2020 Apr 22;35:100684. doi: 10.1016/j.nmni.2020.100684. eCollection 2020 May. PMID 32322397
- [Background] Guzzo CA, Furtek CI, Porras AG, Chen C, Tipping R, Clineschmidt CM, Sciberras DG, Hsieh JY, Lasseter KC. Safety, tolerability, and pharmacokinetics of escalating high doses of ivermectin in healthy adult subjects. J Clin Pharmacol. 2002 Oct;42(10):1122-33. doi: 10.1177/009127002401382731. PMID 12362927
- [Background] Schmith VD, Zhou JJ, Lohmer LRL. The Approved Dose of Ivermectin Alone is not the Ideal Dose for the Treatment of COVID-19. Clin Pharmacol Ther. 2020 Oct;108(4):762-765. doi: 10.1002/cpt.1889. Epub 2020 Jun 7. PMID 32378737
- [Background] Rizzo E. Ivermectin, antiviral properties and COVID-19: a possible new mechanism of action. Naunyn Schmiedebergs Arch Pharmacol. 2020 Jul;393(7):1153-1156. doi: 10.1007/s00210-020-01902-5. Epub 2020 May 27. PMID 32462282
- [Background] Caly L, Druce JD, Catton MG, Jans DA, Wagstaff KM. The FDA-approved drug ivermectin inhibits the replication of SARS-CoV-2 in vitro. Antiviral Res. 2020 Jun;178:104787. doi: 10.1016/j.antiviral.2020.104787. Epub 2020 Apr 3. PMID 32251768
- [Background] Sharun K, Dhama K, Patel SK, Pathak M, Tiwari R, Singh BR, Sah R, Bonilla-Aldana DK, Rodriguez-Morales AJ, Leblebicioglu H. Ivermectin, a new candidate therapeutic against SARS-CoV-2/COVID-19. Ann Clin Microbiol Antimicrob. 2020 May 30;19(1):23. doi: 10.1186/s12941-020-00368-w. No abstract available. PMID 32473642
- [Background] Simsek Yavuz S, Unal S. Antiviral treatment of COVID-19. Turk J Med Sci. 2020 Apr 21;50(SI-1):611-619. doi: 10.3906/sag-2004-145. PMID 32293834
- [Background] Bray M, Rayner C, Noel F, Jans D, Wagstaff K. Ivermectin and COVID-19: A report in Antiviral Research, widespread interest, an FDA warning, two letters to the editor and the authors' responses. Antiviral Res. 2020 Jun;178:104805. doi: 10.1016/j.antiviral.2020.104805. Epub 2020 Apr 21. No abstract available. PMID 32330482
- [Background] Chaccour C, Hammann F, Ramon-Garcia S, Rabinovich NR. Ivermectin and COVID-19: Keeping Rigor in Times of Urgency. Am J Trop Med Hyg. 2020 Jun;102(6):1156-1157. doi: 10.4269/ajtmh.20-0271. No abstract available. PMID 32314704
- [Background] Patri A, Fabbrocini G. Hydroxychloroquine and ivermectin: A synergistic combination for COVID-19 chemoprophylaxis and treatment? J Am Acad Dermatol. 2020 Jun;82(6):e221. doi: 10.1016/j.jaad.2020.04.017. Epub 2020 Apr 10. No abstract available. PMID 32283237
- [Background] Badhan R, Zakaria Z, Olafuyi O. The Repurposing of Ivermectin for Malaria: A Prospective Pharmacokinetics-Based Virtual Clinical Trials Assessment of Dosing Regimen Options. J Pharm Sci. 2018 Aug;107(8):2236-2250. doi: 10.1016/j.xphs.2018.03.026. Epub 2018 Apr 5. PMID 29626533
- [Background] Aroke D, Tchouakam DN, Awungia AT, Mapoh SY, Ngassa SN, Kadia BM. Ivermectin induced Steven-Johnsons syndrome: case report. BMC Res Notes. 2017 May 8;10(1):179. doi: 10.1186/s13104-017-2500-5. PMID 28482929
- [Background] Alout H, Foy BD. Ivermectin: a complimentary weapon against the spread of malaria? Expert Rev Anti Infect Ther. 2017 Mar;15(3):231-240. doi: 10.1080/14787210.2017.1271713. Epub 2016 Dec 29. PMID 27960597
- [Background] Chosidow A, Gendrel D. [Safety of oral ivermectin in children]. Arch Pediatr. 2016 Feb;23(2):204-9. doi: 10.1016/j.arcped.2015.11.002. Epub 2015 Dec 14. French. PMID 26697814
- [Background] Foletto VR, Vanz F, Gazarini L, Stern CA, Tonussi CR. Efficacy and security of ivermectin given orally to rats naturally infected with Syphacia spp., Giardia spp. and Hymenolepis nana. Lab Anim. 2015 Jul;49(3):196-200. doi: 10.1177/0023677214562850. Epub 2014 Dec 5. PMID 25480657
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- See also: SARS-CoV-2 Ivermectin Navarra-ISGlobal Trial (SAINT) — https://www.isglobal.org/healthisglobal/-/custom-blog-portlet/ivermectin-and-covid-19-how-a-flawed-database-shaped-the-covid-19-response-of-several-latin-american-countries/2877257/0